CLINICAL TRIAL: NCT00640133
Title: Controlled Trial of Deep Brain Stimulation for Obsessive-Compulsive Disorder
Brief Title: Effectiveness of Deep Brain Stimulation for Treating People With Treatment Resistant Obsessive-Compulsive Disorder
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Benjamin Greenberg, Professor, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01MH076179 (NIH); U01MH076179 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation; Treatment Refractory; Ventral Internal Capsule/Ventral Striatum; Neurosurgery; Neuroimaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Implantable Neurostimulators

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active DBS (Active Comparator): Participants will receive deep brain stimulation.
  Interventions: Device: Active DBS
- Sham DBS (Sham Comparator): Participants will receive sham deep brain stimulation for several months and then active deep brain stimulation thereafter.
  Interventions: Device: Active DBS; Device: Sham DBS

INTERVENTIONS:
Device: Active DBS — In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will adjust the settings of the electrical stimulation to optimize treatment for each participant. After a post-operative rest, participants will receive immediate DBS treatment throughout.
  Other Names: Activa Deep Brain Stimulation System (Medtronic, Inc.); Implantable Neurostimulator (INS)
Device: Sham DBS — In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months. Afterwards, all participants will receive open-label long-term DBS.
  Other Names: Activa Deep Brain Stimulation System (Medtronic, Inc.); Implantable Neurostimulator (INS)
  Arms: Sham DBS

SUMMARY:
This study will evaluate the safety and effectiveness of deep brain stimulation in treating people with severe and otherwise treatment-resistant obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a chronic and debilitating illness that affects between 2% and 3% of adults in the United States. People with OCD often experience persistent unwanted thoughts and carry out ritual-like behaviors to rid themselves of these obsessive thoughts. Additionally, OCD symptoms are usually tied with feelings of intense anxiety and functional impairment, making it important for people with OCD to seek effective treatment. Although there are currently many treatment options for OCD, including psychotherapy and medications such as serotonin reuptake inhibitors, between 40% and 60% of people with OCD only partially respond or do not respond at all to these treatment methods. Given the large percentage of people who do not respond to aggressive conventional treatments, alternative options are necessary for people with treatment-resistant OCD. Deep brain stimulation (DBS) is a procedure that involves the use of thin wires to carry electric current to parts of the brain associated with producing OCD symptoms. DBS has been effectively and safely used to treat movement disorders, such as Parkinson's disease, and may be beneficial in reducing OCD symptom severity. This study will evaluate the safety and effectiveness of DBS in treating people with severe and otherwise treatment-resistant OCD.

Study participation through follow-up will last 4 years. Participants will be allowed to remain on any pre-surgical medications or behavioral therapy programs throughout the study. Before surgery, all participants will undergo a 3- to 4-day series of initial tests and examinations that will include a physical and neurological examination; blood and urine screening tests; an electrocardiogram (EKG); an electroencephalography (EEG); and detailed psychological testing, including tests of perception, learning, and memory. The EEGs may be performed again after surgery to measure potential changes in brain electrical activity due to DBS.

On the day of the surgery, participants will take a low dose of anxiety medication, have a metal frame fixed to their heads for support during surgery, and undergo a magnetic resonance imaging (MRI) scan to determine where to place the stimulating wires. After being injected with a local anesthetic, participants will undergo the first part of the operation, which will involve the implantation of neurostimulators in the ventral caudate/ventral striatum brain region. For the second part of the operation, after participants are administered general anesthesia, they will have the implantable neurostimulators (INSs) placed in their chests and the connecting wires to the brain placed under their skin. The entire surgical procedure will take 3 to 4 hours, with a 1- to 2-day post-operative hospital stay for recovery. During the post-operative stay, participants will undergo x-rays and a computed tomography (CT) scan of the head.

Two to 3 weeks after surgery, participants will be divided randomly into either a group that receives DBS immediately or a group that first receives sham DBS and then active DBS after 3 months. The level of stimulation will be adjusted individually and on the basis of each participant's response to the stimulation. Participants will complete rating forms, a clinical evaluation, and a check of the stimulators every month for the first 3 months, then at least every 3 months for the rest of the year, and then every 6 months for the remaining years of the study. On the Year 1 visit, participants will repeat the baseline detailed psychological testing. Periodically throughout the 4-year study, staff will contact participants by phone to ask about OCD symptoms, mood, anxiety, and possible side effects. Also throughout the study, participants will need to have the INSs replaced every 5 to 16 months on average.

Participants will also be invited to participate in a related study that involves positron emission tomography (PET) scanning to determine how the stimulation changes activity in the brain. Participation in the separate PET study is optional and will not affect current study participation.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive-compulsive disorder (OCD), diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV)
* Presence of disabling severity, as assessed by a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 30
* Impaired functioning, indicated by a Global Assessment of Functioning (GAF) score of 45 or less
* Documented highly treatment refractory illness; the documentation must demonstrate persistence of severe symptoms and impairment for 5 or more years despite at least three first-line and two second-line treatments, as follows:

  1. at least three adequate trials of, or documented intolerance to, different serotonin transporter inhibitors (e.g., fluoxetine, sertraline, fluvoxamine, paroxetine, citalopram, escitalopram, clomipramine) for at least 3 months at the maximum tolerated dose. These trials may include any of the agents above, but must include an adequate course of clomipramine, either alone or in combination with a more selective serotonin transporter inhibitor;
  2. augmentation of one of the selective serotonin transporter inhibitors with clomipramine, and a neuroleptic (each for at least 2 weeks); and
  3. adequate behavior therapy (more than 20 sessions of exposure and response prevention by a therapist with substantial expertise in OCD treatment as determined by the investigators) with at least one of these trials and tried in combination with medication therapy
* Either drug free or on a stable drug regimen for at least 6 weeks before study entry
* General good overall health
* If possible, has a family member or significant other who sees the participant regularly, can communicate with the study team as needed, and, if necessary, can attend study visits
* Local referring psychiatrist willing to provide ongoing care during and after the trial, to work closely with the research team, and to agree that the study psychiatrist will prescribe medications during the 3-month masked phase
* Platelet count greater than 125,000 per cubic millimeter and a prothrombin time and partial thromboplastin time within normal limits

Exclusion Criteria:

* Current or past psychotic disorder
* Full-scale IQ below 75 on the Wechsler Abbreviated Scale of Intelligence (WASI), or cognitive impairment that would affect a participant's ability to give informed consent or provide interview or self-report data reliably, as determined by the Consent Monitor and the site psychiatrist.
* A clinical history of bipolar mood disorder
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than a tic disorder
* Any clinically significant abnormality on preoperative MRI
* Any labeled DBS contraindication, inability to undergo presurgical MRI (e.g., cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac risk factors, or other medical risk factors for surgery
* Current or unstable remitted substance abuse or dependence
* Positive urine toxicology screen for substance abuse
* Pregnant and/or woman of childbearing age not using effective forms of birth control
* Clinical history of severe personality disorder
* An inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death
* Current diagnosis of body dysmorphic disorder
* Evidence of dementia of other significant cognitive impairment on neuropsychological evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2018-05-24 (Actual); Study Completion 2024-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Greenberg, MD, PhD, Principal Investigator — Butler Hospital/Brown University
Locations (9):
- United States (9):
  - Kaiser Permanente Redwood City Hospital, Redwood City, California
  - George Washington University Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Greenberg BD, Malone DA, Friehs GM, Rezai AR, Kubu CS, Malloy PF, Salloway SP, Okun MS, Goodman WK, Rasmussen SA. Three-year outcomes in deep brain stimulation for highly resistant obsessive-compulsive disorder. Neuropsychopharmacology. 2006 Nov;31(11):2384-93. doi: 10.1038/sj.npp.1301165. Epub 2006 Jul 19. PMID 16855529
- [Result] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Result] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Result] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Result] Kanter, J. W., Rusch, L. C., Busch, A. M., & Sedivy, S. K. (2009). Validation of the behavioral activation for depression scale (BADS) in a community sample with elevated depressive symptoms. Journal of Psychopathology and Behavioral Assessment, 31, 36-42.
- [Result] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Result] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Result] American Psychiatric Association. (2000). Diagnostic and statistical manual of mental disorders, (4th ed., text revision). Washington, DC: American Psychiatric Association.
- [Derived] McLaughlin NC, Didie ER, Machado AG, Haber SN, Eskandar EN, Greenberg BD. Improvements in anorexia symptoms after deep brain stimulation for intractable obsessive-compulsive disorder. Biol Psychiatry. 2013 May 1;73(9):e29-31. doi: 10.1016/j.biopsych.2012.09.015. Epub 2012 Nov 3. No abstract available. PMID 23128051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is a parallel controlled design. Patients (n=27) were assigned to a condition by site & gender via urn randomization to receive three months of double-masked sham or double-masked active DBS. After 3 months, all patients received open-label active DBS. 12 patients were in the sham group while 15 patients received active DBS immediately.
Groups:
- Sham DBS: Participants will receive sham deep brain stimulation for three months and then active deep brain stimulation thereafter.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months.
  Active DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will adjust the settings of the electrical stimulation to optimize treatment for each participant. After a post-operative rest, participants will receive immediate DBS treatment throughout.
Period: Randomization Phase (Baseline-Month 3)
Arm/Group | Active DBS | Sham DBS
Started | 15 | 12
Completed | 15 | 12
Not Completed | 0 | 0
Period: Open Label Phase (Month 4-12)
Arm/Group | Active DBS | Sham DBS
Started | 27 | 0
Completed | 24 | 0
Not Completed | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham DBS: Participants will receive sham deep brain stimulation for 3 months and then active deep brain stimulation thereafter.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months. Afterwards, all participants will receive open-label long-term DBS.
- Total: Total of all reporting groups
Arm/Group | Active DBS | Sham DBS | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.9) | 35.1 (10.5) | 39.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — All patients must receive follow-up and DBS programming at one of the 8 collaborative study sites. If a patient is not located within 2 hours of a study site, FDA-approval must be granted for additional study sites.
  Participants
    United States | 15 | 12 | 27
Yale-Brown Obsessive-Compulsive Scale (YBOCS) [Mean (Standard Deviation); unit: units on a scale] — The Yale-Brown Obsessive-Compulsive Scale (YBOCS) is a 10 question evaluator-administered measure assessing the severity of obsessions and compulsions over the past week (each of the 10 items are rated 0-4; 4 being the most severe). Total scores are summed and range from 0-40. Higher scores for obsessions, compulsions and total score indicate more severe symptoms over the past week.
  units on a scale | 33.3 (2.3) | 33.5 (2.3) | 33.5 (2.3)
Global Assessment of Functioning (GAF) [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Functioning (GAF) scale is a numeric scale (0 through 100) used to rate the social, occupational, and psychological overall functioning during the week of poorest functioning in the past month. Higher scores indicate a higher level of functioning, while low scores indicate impaired global functioning.
  units on a scale | 37.0 (6.8) | 41.6 (2.9) | 39.0 (5.8)
Social and Occupational Functioning Assessment Scale (SOFAS) [Mean (Standard Deviation); unit: units on a scale] — The Social and Occupational Functioning Assessment (SOFAS) is a numeric scale (0 through 100) used to rate the social, occupational, and psychological functioning during the week of poorest functioning in the past month. Higher scores indicate higher levels of social and occupational functioning, while low scores represent social and occupational impairment.
  units on a scale | 38.5 (8.0) | 41.5 (3.9) | 39.9 (6.6)
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-administered measure to assess the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning. We used the 16-item short form with total scores ranging from 16-80. Higher scores indicate greater satisfaction experienced during the past week.
  units on a scale | 36.7 (9.8) | 37.6 (7.7) | 37.5 (8.8)
The Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Asberg Depression Rating Scale (MADRS) is an interviewer-administered measure assessing the ten symptoms of depression most sensitive to change. Apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts are assessed and total scores range from 0-60 with higher scores representing the presence of more severe depression over the past week.
  units on a scale | 25.6 (7.6) | 19.9 (13.5) | 22.7 (10.8)
Hamilton Anxiety Rating Scale (HARS) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Anxiety Rating Scale (HARS) is a 14-item test measuring the severity of anxiety symptoms. It provides measures of overall anxiety, psychic anxiety (mental agitation and psychological distress), and somatic anxiety (physical complaints related to anxiety); total scores range from 0-56. Higher scores indicate higher levels of anxiety over the past week.
  units on a scale | 19.3 (7.2) | 16.7 (10.3) | 17.6 (8.9)
Behavioral Activation Scale for Depression (BADS) [Mean (Standard Deviation); unit: units on a scale] — The Behavioral Activation for Depression Scale (BADS) is a 29-item scale that measures the role of aversive controlling stimuli and escape and avoidance behavior in depression, specifically when and how participants become more activated over the course of treatment. Total scores range from 29-203 and lower scores indicate higher levels of escape and avoidance behavior from depression in the past week.
  units on a scale | 67.5 (25.4) | 72.0 (17.6) | 69.7 (21.8)
Hamilton Depression Rating Scale (HDRS) [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale (HDRS) measures the severity of depressive symptoms in adults. The evaluator-administered ratings measure depressed mood, guilt, suicide, insomnia, work/activities, retardation, agitation, psychic and somatic anxiety, genital symptoms, hypochondriasis, and insight during the past week. Total scores range from 0-72 and higher scores indicate the presence of more severe depression over the past week. Note: this measure was only administered at baseline and month-3.
  units on a scale | 29.0 (9.2) | 22.4 (11.3) | 26.1 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive-Compulsive Scale (YBOCS Severity Ratings)
Description: The Yale-Brown Obsessive-Compulsive Scale (YBOCS) is a 10 question evaluator-administered measure assessing the severity of obsessions and compulsions over the past week. Obsession and compulsion severity are evaluated separately (ratings from 0-20 for each category) with total scores ranging from 0-40. Higher scores for obsessions, compulsions and total score indicate more severe symptoms over the past week.
Time Frame: YBOCS total score observed means at month-12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham DBS: Participants will receive sham deep brain stimulation for several months and then active deep brain stimulation thereafter.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months.
  Afterwards, all participants will receive open-label long-term DBS.
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 12 | 12
units on a scale | 20.5 (10.6) | 20.9 (7.0)

2. Primary Outcome: Global Assessment of Functioning Scale (GAF)
Description: A numeric scale (0 through 100) used to rate the social, occupational, and psychological overall functioning during the week of poorest functioning in the past month. Higher scores indicate a higher level of functioning, while low scores indicate impaired global functioning.
Time Frame: GAF score observed means at month-12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham DBS: Participants will receive sham deep brain stimulation for several months and then active deep brain stimulation thereafter.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months.
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 12 | 12
units on a scale | 54.8 (16.5) | 53.7 (8.2)

3. Primary Outcome: Social and Occupational Functioning Assessment Scale (SOFAS)
Description: A numeric scale (0 through 100) used to rate the social, occupational, and psychological functioning during the week of poorest functioning in the past month. Higher scores indicate higher levels of social and occupational functioning, while low scores represent social and occupational impairment.
Time Frame: SOFAS score observed means at month-12 time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 12 | 12
units on a scale | 55.9 (16.0) | 53.9 (7.1)

4. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is a self-administered measure to assess the degree of enjoyment and satisfaction experienced by participants in various areas of daily functioning. We used the 16-item short form with total scores ranging from 16-80. Higher scores indicate greater satisfaction experienced during the past week.
Time Frame: QLESQ total score observed means at month-12 time point.
Population: In total, 4 participants receiving active DBS did not complete Q-LES-Q ratings at month 12; 3 participants exited the protocol before the month-12 endpoint and 1 participant had incomplete Q-LES-Q data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 11 | 12
units on a scale | 39.8 (12.8) | 42.7 (8.4)

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is an interviewer-administered measure assessing the ten symptoms of depression most sensitive to change. Apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts are assessed and total scores range from 0-60 with higher scores representing the presence of more severe depression over the past week.
  interviewer-administered measure assessing
Time Frame: MADRS total score observed means at month-12 time point.
Population: In total, 4 participants receiving active DBS did not complete MADRS ratings at month 12; 3 participants exited the protocol before the month-12 endpoint and 1 participant had incomplete MADRS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 11 | 12
units on a scale | 17.1 (12.8) | 18.5 (10.1)

6. Secondary Outcome: Hamilton Anxiety Rating Scale (HARS)
Description: Hamilton Anxiety Rating Scale (HARS) is a 14-item test measuring the severity of anxiety symptoms. It provides measures of overall anxiety, psychic anxiety (mental agitation and psychological distress), and somatic anxiety (physical complaints related to anxiety); total scores range from 0-56. Higher scores indicate higher levels of anxiety over the past week.
Time Frame: HARS total score observed means at month-12 time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 12 | 12
units on a scale | 12.6 (8.8) | 15.7 (11.4)

7. Secondary Outcome: Behavioral Activation for Depression Scale (BADS)
Description: The Behavioral Activation for Depression Scale (BADS) is a 29-item scale that measures the role of aversive controlling stimuli and escape and avoidance behavior in depression, specifically when and how participants become more activated over the course of treatment. Total scores range from 29-203 and lower scores indicate higher levels of escape and avoidance behavior from depression in the past week.
Time Frame: Total BADS score observed means at month-12 time point.
Population: In total, 4 participants receiving active DBS did not complete BADS ratings at month 12; 3 participants exited the protocol before the month-12 endpoint and 1 participant had incomplete BADS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 11 | 12
units on a scale | 85.3 (28.9) | 80.3 (22.7)

8. Secondary Outcome: Hamilton Depression Rating Scale (HDRS)
Description: The Hamilton Depression Rating Scale (HDRS) measures the severity of depressive symptoms in adults. The evaluator-administered ratings measure depressed mood, guilt, suicide, insomnia, work/activities, retardation, agitation, psychic and somatic anxiety, genital symptoms, hypochondriasis, and insight during the past week. Total scores range from 0-72 and higher scores indicate the presence of more severe depression over the past week. Note: this measure was only administered at baseline and month-3.
Time Frame: Total HDRS score observed means at month-3 time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham DBS: Participants will receive sham deep brain stimulation for several months and then active deep brain stimulation thereafter.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months.
  Sham DBS: In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will mimic adjusting the settings of the electrical stimulation. After a post-operative rest, participants will receive DBS treatment after a delay of several months. Afterward
Arm/Group | Active DBS | Sham DBS
Number analyzed (Participants) | 15 | 12
units on a scale | 16.8 (9.6) | 19.4 (13.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected beginning after DBS device implantation and continued throughout each patient's participation in the study up to four years post-implantation and up to one year after exiting the protocol.
Arm/Group | Active DBS | Sham DBS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/15 | 1/12
Other Adverse Events (participants affected / at risk) | 10/15 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active DBS (N=15) | Sham DBS (N=12)
Symptom worsening (Nervous system disorders) | 1 (1) | 0 (0) — Mood liability alternating between irritable, anger and sad, worsening to SI hurting self and wanting to die.
Motor effect (fall) (Nervous system disorders) | 1 (1) | 0 (0) — Patient rolled out of bed and hit head. Went to ER, received 6 stitches on scalp.
Periorbital swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient went to ER due to periorbital swelling.
Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — New infection, "boil," developed at implant site and expelled pus and blood.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active DBS (N=15) | Sham DBS (N=12)
Symptom worsening (Nervous system disorders) | 4 (9) | 4 (8) — Including increased anxiety, OCD, depression,
Hypomania (Nervous system disorders) | 1 (1) | 2 (3) — Hypomania also including "elevated mood"
Alcohol-related event (Nervous system disorders) | 1 (2) | 0 (0) — Fight and shoulder pain from drunken fall.
Post-surgical discomfort/pain (Injury, poisoning and procedural complications) | 2 (4) | 1 (1) — Discomfort/pain/numbness after surgery
Infection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Post-surgical infection
Pocket stimulation (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) — Side effect of the device.
GI discomfort/symptoms (Gastrointestinal disorders) | 1 (2) | 3 (4) — GI discomfort including diarrhea, abdominal pain, and bleeding
Headache/migraine (Nervous system disorders) | 1 (3) | 2 (2) — Headache/migraine (including chronic)
Tiredness/severe fatigue (Nervous system disorders) | 2 (3) | 0 (0) — Tiredness up to severe fatigue
Insomnia (Nervous system disorders) | 0 (0) | 1 (2) — Insomnia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT00640133/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT00640133/SAP_000.pdf